CLINICAL TRIAL: NCT00855374
Title: PAR Regulation of Platelet Function in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Heidi Hamm, Professor and Chair of Pharmacology, Vanderbilt University
Other Study IDs: 070474
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Diabetes Mellitus; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Thrombin is the most potent activator of platelets, and platelet activation is a hallmark of thrombosis. Coronary artery disease (CAD) is the major cause of mortality and morbidity in the United States and other industrialized countries, and thrombotic sequelae are the key cause of death in diabetes. The accumulation of thrombin at sites of vascular injury provides one of the major mechanisms of recruiting platelets into a hemostatic plug. Thrombin works by activation of the G protein-coupled protease activated receptors PAR1 and PAR4 on human platelets to initiate signaling cascades leading to increases in [Ca]i, secretion of autocrine activators, trafficking of adhesion molecules to the plasma membrane, and shape change, which all promote platelet aggregation. The thrombin receptors work in a progressive manner, with PAR1 activated at low thrombin concentrations, and PAR4 recruited at higher thrombin concentrations. As direct thrombin inhibitors become widely used in clinical practice, it is important to assess their effects on vascular function. Our hypothesis is that PAR1 and PAR4 do not signal through the same G protein pathways, and that PAR4 is not a strong platelet agonist. To investigate this hypothesis, the investigators will study the G protein pathways downstream of PAR4, and assess ex-vivo platelet responsiveness to thrombin, PAR1, and PAR4 agonist peptides, both in normal human subjects, and along the stages of pathology, from patients with stable angina as well as unstable angina who are undergoing angioplasty. Similarly, the investigators will examine platelet function in patients with metabolic syndrome as well as diabetes, along the continuum from insulin resistance to full-blown disease. These studies will provide deeper insight into the G protein pathways used by PARs. They will elucidate the contribution of PAR receptors to normal platelet function as well as the abnormal platelet activation in thrombotic states. The long term goal is to understand the implications for PAR receptors as therapeutic targets for anti-platelet therapies that may carry less bleeding risk.

DETAILED DESCRIPTION:
Given the known roles of proteases and PARs in coagulation, inflammation, pain, healing and protection, the need for development of a PAR antagonist as a therapeutic agent for treatment of thrombosis, atherosclerosis and inflammation is well-recognized. Thus, blocking PAR action by inhibiting the PAR-G protein interface is an alternative target for blocking downstream consequences of thrombin-mediated cellular activation. Since there are two PARs on human platelets, PAR1 and PAR4, it is critical to define the roles of both receptors in several likely clinical settings where PAR antagonists would be used. In this proposal both the G protein pathways underlying PAR signaling mechanisms as well as their roles in pathologies characterized by activated platelets will be studied in detail. We propose in our grant to investigate the specific roles of individual PARs in mediating the events leading to the multi-stage process of platelet activation and clot formation. The long term goals of these studies are to determine novel PAR-specific anti-platelet therapies. The 2002 estimates of the DHHS suggest that 6.3% of the population of the United States (18.2 Million people) have diabetes, with estimated annual costs of $132 Billion (Centers for Disease Control and Prevention). The complications of coronary artery and of cerebrovascular disease account for up to 65% of deaths in patients with diabetes. The prevalence, complexity and complications of cardiovascular disease are increased in patients with diabetes. This appears related to the frequent association of diabetes and of insulin resistance with traditional risk factors for atherosclerosis. Recent studies by Haffner and other investigators have established the concept of diabetes as a coronary risk equivalent; this is reflected in the guidelines for therapeutic targets set by the ADA, AHA and ACC.

The clinical importance of platelet activation is reflected by the benefits of aspirin and clopidogrel and GPIIbIIIa inhibitors in diabetics. Epidemiologic data demonstrates that the metabolic syndrome is associated with an increased incidence of atherosclerotic events. Type 2 diabetes shares many features in common with the metabolic syndrome, and may represent a precursor condition, Stern described this in the "common soil hypothesis". Hsueh and Law have more recently proposed that the progression of insulin resistance to type 2 diabetes parallels the progression of endothelial dysfunction to atherosclerosis.

These studies were designed to study PAR signaling and G protein activation states in patients with platelet activation in the setting of the continuum of the metabolic syndrome and diabetes mellitus. The degree of platelet activation as determined by assays of platelet reactivity and by the expression of markers of platelet activation will be correlated with the changes in PAR signaling. These studies will provide a comprehensive assessment of platelet activation in the setting of the metabolic syndrome, and will compare the extent of activation in this setting with that in a group of contemporaneously studied patients with diabetes mellitus. Finally, the influence of the direct thrombin inhibitor, bivalirudin on platelet activation and signaling will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18, Sex: male and female.
* Patients who undergo clinically indicated coronary angiography and/or PCI. Patients in Group 1 (elective PCI) include those presented with stable angina (ACC definition for stable angina).
* Coronary angiography reveals severe stenosis (>70%) that requires PCI.
* Patients in Group 2 (elective PCI in subjects with diabetes) include those who present with stable angina, or with findings on non-invasive testing (exercise or pharmacologic stimulation with imaging by nuclear perfusion imaging or stress echocardiography) in whom coronary angiography reveals severe stenosis (>70%) that requires PCI.
* Patients in Group 2 (ACS) include those presented with unstable angina or non-ST elevation myocardial infarction (as defined by the ACC).
* Coronary angiography reveals severe stenosis (>70%) that requires PCI.

Exclusion Criteria:

* Significant left main coronary artery disease.
* Severely impaired left ventricular systolic function (EF<35%).
* Prior treatment with enoxaparin, Bivalirudin (or other thrombin inhibitors), Warfarin, or thrombolytic agents <48 hours. Prior history of myocardial infarction (<6 weeks).
* Prior history of stroke (<6 weeks).
* Prior history of coronary intervention (<6 weeks).
* History of HIV/AIDS.
* The patients will be identified in the following manner:
* All subjects will be picked from a pool of patients diagnosed with stable angina and diabetes from the Vanderbilt Page-Campbell Heart Institute at Vanderbilt University Medical Center and undergo a complete history and physical examination. Patients with acute coronary syndrome will be referred from the acute cardiology patient service at Vanderbilt University Medical Center.
* Subjects with hematologic, renal (creatinine > 2.0 mg/dl), hepatic, inflammatory, and neoplastic disorders, and those who sustained a recent (< 1 month) myocardial infarction, ACS, or stroke will be excluded.
* Patients who used nonsteroidal anti-inflammatory drugs, corticosteroids, or hormone replacement therapy will also be excluded.
* Pregnancy will be excluded in women of child bearing potential by measurement of urine ß-HCG (it is standard of care to determine if a woman is pregnant prior to elective PCI and will be screened as part of their PHI).
* For healthy volunteers, pregnancy will be excluded per verbal report.
* Data will be collected regarding patient demographics including height and weight, abdominal circumference, blood pressure, comorbid medical conditions, triglycerides, HDL, fasting glucose and medication use (including prescription of antithrombotic agents, ACE inhibitors, angiotensin receptor blockers, beta blockers, calcium channel antagonists and HMG-CoA inhibitors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic patients in the Vanderbilt General Clinical Research Center
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2008-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi E Hamm, Ph.D., Principal Investigator — Vanderbilt University Medical Center, Pharmacology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States